CLINICAL TRIAL: NCT02155153
Title: The Effect of Gum Chewing on the Duration of Postoperative Ileus and Total Length of Hospital Stay After Reversal of Ileostomy
Brief Title: Role of Chewing Gum in Reducing Post Operative Ileus After Reversal of Ileostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Services Hospital, Lahore (Other Government)
Responsible Party: Principal Investigator, Dr. SamiUllah, Medical Officer, Services Hospital, Lahore
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: cg1
Record Dates: First submitted 2014-06-01; First posted 2014-06-04 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Postoperative Ileus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar Free Chewing Gum (Experimental): All patients receiving sugar free gum
  Interventions: Other: Sugar Free Chewing Gum
- Control (No Intervention): Patients receiving no intervention

INTERVENTIONS:
Other: Sugar Free Chewing Gum — 'Extra' sugar free gum will be used as an intervention. Patients will be required to chew a gum for 30 min at intervals of 6 hours for first 48 hours post operatively or until they pass flatus.
  Other Names: 'Extra' Sugar Free Gum
  Arms: Sugar Free Chewing Gum

SUMMARY:
Postoperative ileus is generally referred to as the transient impairment of bowel motility after abdominal or other surgery and diagnosed by postoperative abdominal pain vomiting constipation and distension.

The potential complications of prolonged POI include increased postoperative pain, increased nausea and vomiting, pulmonary complications, poor wound healing, delay in resuming oral intake, delay in postoperative mobilization, prolonged hospitalization, and increased health-care costs. The estimated economic impact of POI in the United States is $7.5 billion per year, excluding the expenses of work loss.

In view of these complications and economic burden a number of pharmacologic and non-pharmacologic strategies have been adopted by the doctors all over the world to reduce the burden of postoperative ileus.These programs involve transverse or curved surgical incisions, removal of nasogastric tubes at the end of anesthesia, intraoperative and postoperative analgesia, early postoperative feeding, mobilization, and gum chewing.

The use of gum chewing has emerged as a new and simple modality for decreasing POI. And reviews have concluded that there is consistent benefit for patients from gum chewing after the intestinal surgery; colonic surgery and gynecological surgery.

This study is based on the hypothesis that postoperative gum chewing is beneficial in prevention of postoperative ileus after reversal of ileostomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either gender with age ranging from 15 to 60 years.
2. Patients whose ileostomies were made for typhoid or tuberculous perforation
3. Patients with no distal obstruction on loopogram.

Exclusion Criteria:

- 1. Patients with age less than 15 years and greater than 60. 2. Patients having co-morbid factors such as diabetes and ischemic heart disease.

3. Patients whose ileostomy was made for any condition other than typhoid or tuberculosis.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
passage of flatus | within 48 hours after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Mahmood Ayyaz, FCPS FACS, Study Director — Professor of Surgery
Locations (1):
- Services hospital lahore, Lahore, Punjab Province, Pakistan